CLINICAL TRIAL: NCT00847379
Title: A Phase 2B Extension Study of PTC124 in Subjects With Nonsense-Mutation-Mediated Duchenne and Becker Muscular Dystrophy
Brief Title: Phase 2B Extension Study of Ataluren (PTC124) in Duchenne/Becker Muscular Dystrophy (DMD/BMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-007e-DMD
Record Dates: First submitted 2009-02-16; First posted 2009-02-19 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Becker muscular dystrophy; Nonsense mutation; Premature stop codon; DMD; BMD; Ataluren; PTC124
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overall Participants: High-Dose Ataluren (Experimental): All participants will receive ataluren suspension orally three times a day (TID), 20 mg/kg at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for up to 96 weeks in this study. Any participant who was receiving a reduced dose of ataluren at the end of treatment visit in study PTC124-GD-007-DMD, will be initiated ataluren therapy in this extension study at the 5-, 5-, and 10-mg/kg dose level; dose will be increased to 10, 10, and 20 mg/kg at Week 6 and to 20, 20, and 40 mg/kg at Week 12, if the preceding dose level is well tolerated.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren oral powder for suspension will be administered as per dose and schedule specified in the arm.
  Other Names: PTC124

SUMMARY:
Duchenne/Becker muscular dystrophy (DMD/BMD) is a genetic disorder that develops in boys. It is caused by a mutation in the gene for dystrophin, a protein that is important for maintaining normal muscle structure and function. Loss of dystrophin causes muscle fragility that leads to weakness and loss of walking ability during childhood and teenage years. A specific type of mutation, called a nonsense (premature stop codon) mutation is the cause of DMD/BMD in approximately 10-15% of boys with the disease. Ataluren (PTC124) is an orally delivered, investigational drug that has the potential to overcome the effects of the nonsense mutation. This study is a Phase 2b extension trial that will evaluate the long-term safety of ataluren (PTC124) in boys with nonsense mutation DMD/BMD, as determined by adverse events and laboratory abnormalities. The study will also assess changes in walking, muscle function, and other important clinical and laboratory measures.

DETAILED DESCRIPTION:
This is a Phase 2b, international, multicenter, open-label extension study for participants who successfully completed blinded study drug in Study 007. This extension study will evaluate the long-term administration of ataluren administered 3 times per day (TID) at morning, midday, and evening doses of 20, 20, and 40 milligrams/kilogram (mg/kg), respectively, in participants with nonsense mutation Duchenne/Becker muscular dystrophy (nmDBMD).

ELIGIBILITY:
Inclusion Criteria:

* Completion of blinded study drug treatment in the previous Phase 2b study (PTC124-GD-007-DMD).
* Ability to provide written informed consent (parental/guardian consent if applicable)/assent (if less than [<]18 years of age).
* In participants who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during PTC124 administration and the 6-week follow up period.
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions.

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug (Litesse® UltraTM [refined polydextrose], polyethylene glycol 3350, Lutrol® micro F127 [poloxamer 407], mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, Cab-O-Sil® M5P [colloidal silica], magnesium stearate).
* Ongoing participation in any other therapeutic clinical trial.
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow up would be completed, or could impair the assessment of study results.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-01-31 (Actual); Primary Completion 2010-05-24 (Actual); Study Completion 2010-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leone Atkinson, M.D., Ph.D., Study Director — PTC Therapeutics
Locations (37):
- United States (15):
  - University of California - Davis, Sacramento, California
  - Department of Rehabilitation, The Children's Hospital, Aurora, Colorado
  - Child Neurology Center of NW Florida, Gulf Breeze, Florida
  - University of Iowa Children's Hospital, Division of Child Neurology, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriners Hospital for Children-Portland, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Southwestern University, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - The Royal Children's Hospital, Parkville, Victoria
  - The Children's Hospital at Westmead, Westmead
- UZ Leuven, Leuven, Belgium
- Canada (3):
  - Alberta Children's Hospital, London, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - British Colombia Children's Hopsital, Vancouver
- France (3):
  - Hopital d'Enfants CHU Timone, Marseille
  - Laboratoire d'Exploration Fonctionnelles, Nantes
  - Groupe Hospitalier Pitie-Salpetriere, Institut de Myologie, Paris
- Germany (2):
  - University of Essen - Clinic for Children, Essen
  - University Hospital, Freiburg im Breisgau
- Hadassah University Hopspital, Jerusalem, Israel
- Italy (3):
  - Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Ospedale Pediatrico Bambino Gesu, Roma
  - U.O. Complessa di Neuropsichiatria Infantile-Policlinico A. Gemelli-Universita Cattolica, Roma
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario La Fe, Valencia
- Sweden (2):
  - Queen Silvia Children's Hospital, Gothenburg
  - Astrid Lindgren Pediatric Hospital, Stockholm
- United Kingdom (3):
  - UCL Instititute of Child Health, Dubowitz, London
  - University of Newcastle, Newcastle upon Tyne
  - Robert Jones & Agnes Hunt Orthopaedic Hospital, Oswestry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirawat S, Welch EM, Elfring GL, Northcutt VJ, Paushkin S, Hwang S, Leonard EM, Almstead NG, Ju W, Peltz SW, Miller LL. Safety, tolerability, and pharmacokinetics of PTC124, a nonaminoglycoside nonsense mutation suppressor, following single- and multiple-dose administration to healthy male and female adult volunteers. J Clin Pharmacol. 2007 Apr;47(4):430-44. doi: 10.1177/0091270006297140. PMID 17389552
- [Background] Welch EM, Barton ER, Zhuo J, Tomizawa Y, Friesen WJ, Trifillis P, Paushkin S, Patel M, Trotta CR, Hwang S, Wilde RG, Karp G, Takasugi J, Chen G, Jones S, Ren H, Moon YC, Corson D, Turpoff AA, Campbell JA, Conn MM, Khan A, Almstead NG, Hedrick J, Mollin A, Risher N, Weetall M, Yeh S, Branstrom AA, Colacino JM, Babiak J, Ju WD, Hirawat S, Northcutt VJ, Miller LL, Spatrick P, He F, Kawana M, Feng H, Jacobson A, Peltz SW, Sweeney HL. PTC124 targets genetic disorders caused by nonsense mutations. Nature. 2007 May 3;447(7140):87-91. doi: 10.1038/nature05756. Epub 2007 Apr 22. PMID 17450125
- See also: Sponsor's web site — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 173 participants were screened for eligibility to enter this extension study after completing the 48-week double-blind study PTC124-GD-007-DMD (NCT00592553). All participants met entry criteria and enrolled in this study.
Pre-assignment Details: Participants were categorized by the treatment group to which they had been randomly assigned in Study PTC124-GD-007-DMD (NCT00592553).
Groups:
- High-Dose Ataluren/High-Dose Ataluren: Participants who were randomized to receive high-dose ataluren in study PTC124-GD-007-DMD, continued to receive ataluren suspension orally 3 times a day (TID), 20 milligrams/kilogram (mg/kg) at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for up to 96 weeks in this study. Any participant who was receiving a reduced dose of ataluren at the end of treatment visit (Week 48) in study PTC124-GD-007-DMD, was initiated ataluren therapy in this extension study at the 5-, 5-, and 10-mg/kg dose level; dose was increased to 10, 10, and 20 mg/kg at Week 6 and to 20, 20, and 40 mg/kg at Week 12, if the preceding dose level was well tolerated.
- Low-Dose Ataluren/High-Dose Ataluren: Participants who were randomized to receive low-dose ataluren in study PTC124-GD-007-DMD, received ataluren suspension orally TID, 20 mg/kg at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for up to 96 weeks in this study. Any participant who was receiving a reduced dose of ataluren at the end of treatment visit in study PTC124-GD-007-DMD, was initiated ataluren therapy in this extension study at the 5-, 5-, and 10-mg/kg dose level; dose was increased to 10, 10, and 20 mg/kg at Week 6 and to 20, 20, and 40 mg/kg at Week 12, if the preceding dose level was well tolerated.
- Placebo/High-Dose Ataluren: Participants who were randomized to receive placebo in study PTC124-GD-007-DMD, received ataluren suspension orally TID, 20 mg/kg at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for up to 96 weeks in this study. Any participant who was receiving a reduced dose of placebo at the end of treatment visit in study PTC124-GD-007-DMD, was initiated ataluren therapy in this extension study at the 5-, 5-, and 10-mg/kg dose level; dose was increased to 10, 10, and 20 mg/kg at Week 6 and to 20, 20, and 40 mg/kg at Week 12, if the preceding dose level was well tolerated.
Period: Overall Study
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren
Started | 59 | 57 | 57
As-treated Population (All participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e.) | 59 | 57 | 57
Completed | 0 | 0 | 0
Not Completed | 59 | 57 | 57
Not completed — Study terminated by Sponsor | 59 | 57 | 57

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who completed Study 007 and received greater than or equal to (≥) 1 dose of ataluren in Study 007e.
Groups:
- High-Dose Ataluren/High-Dose Ataluren: Participants who were randomized to receive high-dose ataluren in study PTC124-GD-007-DMD, continued to receive ataluren suspension orally TID, 20 mg/kg at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for up to 96 weeks in this study. Any participant who was receiving a reduced dose of ataluren at the end of treatment visit in study PTC124-GD-007-DMD, was initiated ataluren therapy in this extension study at the 5-, 5-, and 10-mg/kg dose level; dose was increased to 10, 10, and 20 mg/kg at Week 6 and to 20, 20, and 40 mg/kg at Week 12, if the preceding dose level was well tolerated.
- Total: Total of all reporting groups
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Total
Number analyzed (Participants) | 59 | 57 | 57 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (2.53) | 9.7 (2.89) | 9.3 (2.28) | 9.5 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 59 | 57 | 57 | 173

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of an AE was classified as: mild (does not interfere with usual function), moderate (interferes to some extent with usual function) and severe (interferes significantly with usual function). Drug-related AEs: AEs with a possible or probable relationship to study drug. Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention. TEAE: AE that occurred or worsened in the period extending from first dose of study drug in this study to 6 weeks after last dose of study drug in this study. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Week 48 of Study 007) up to Week 102
Population: As-treated population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Participants: High-Dose Ataluren: All participants received ataluren suspension orally TID, 20 mg/kg at morning, 20 mg/kg at midday, and 40 mg/kg at evening (total daily dose 80 mg/kg) for up to 96 weeks in this study. Any participant who was receiving a reduced dose of ataluren at the end of treatment visit in study PTC124-GD-007-DMD, was initiated ataluren therapy in this extension study at the 5-, 5-, and 10-mg/kg dose level; dose was increased to 10, 10, and 20 mg/kg at Week 6 and to 20, 20, and 40 mg/kg at Week 12, if the preceding dose level was well tolerated.
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 59 | 57 | 57 | 173
Participants
  Any AEs | 52 | 49 | 48 | 149
  Drug-related AEs | 10 | 10 | 22 | 42
  Serious AEs | 0 | 1 | 2 | 3
  Mild AEs | 34 | 23 | 26 | 83
  Moderate AEs | 13 | 22 | 19 | 54
  Severe AEs | 5 | 4 | 3 | 12

2. Primary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Laboratory parameters tests included hematology, biochemistry assay (hepatic, renal, and serum electrolyte values), adrenal assays, and urinalysis. Clinical significance was defined as per investigator's judgement.
Time Frame: Baseline (Week 48 of Study 007) up to Week 102
Population: As-treated population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 59 | 57 | 57 | 173
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Week 60
Description: The 6MWD test was performed in a 30 meters long flat corridor, where the participant was instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: Ambulatory 007e population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e, and had sufficient baseline and on-treatment data in Study 007e to assess measure of interest, excluding participants who had lost all independent ambulation. 'Number analyzed'=participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
meters
  Baseline | 351.60 (130.312) | 375.95 (98.976) | 356.25 (109.369) | 361.11 (113.760)
  Change at Week 60: number analyzed (Participants) | 46 | 46 | 47 | 139
  Change at Week 60 | -17.23 (39.608) | -10.50 (41.390) | -7.06 (50.121) | -11.56 (43.881)

4. Secondary Outcome: Change From Baseline in Mean Activity Period/Day/Visit at Week 60, as Assessed by Step Activity Monitoring (SAM)
Description: The SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). Mean activity period/day/visit was computed for each participant. For each day, an active period was defined as the first time after 3:00 AM that greater than (>) 2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was less than (<) 50 percent (%) of the mean active period across all days for that participant's visit.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
meters
  Baseline: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline | 759.715 (77.5210) | 742.223 (107.7264) | 747.464 (102.6531) | 750.016 (96.1057)
  Change at Week 60: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60 | 1.946 (61.2247) | 34.283 (88.1587) | -1.866 (93.0531) | 10.991 (82.6356)

5. Secondary Outcome: Change From Baseline in Mean Total Step Count/Day/Visit During the Active Periods at Week 60, as Assessed by SAM
Description: The SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). Mean total step count/day/visit during the active periods was computed for each participant. For each day, an active period was defined as the first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
steps
  Baseline: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline | 4934.575 (2433.230) | 4543.766 (2051.300) | 5175.330 (2307.436) | 4883.613 (2272.108)
  Change at Week 60: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60 | -357.679 (1232.109) | -215.062 (1761.773) | -647.504 (1680.522) | -409.558 (1566.386)

6. Secondary Outcome: Change From Baseline in Mean Total Step Count/Hour During the Active Period at Week 60, as Assessed by SAM
Description: The SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). Mean total step count/hour during the active periods for the days in a visit was computed for each participant. For each day, an active period was defined as the first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
steps
  Baseline: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline | 395.491 (200.7671) | 368.672 (155.6648) | 420.684 (188.9124) | 394.787 (183.0994)
  Change at Week 60: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60 | -27.650 (87.8797) | -34.693 (128.0609) | -54.755 (122.4142) | -39.010 (113.3481)

7. Secondary Outcome: Change From Baseline in Maximum Continuous 10-minute, 20-minute, 30-minute, and 60-minute Total Step Count at Week 60, as Assessed by SAM
Description: SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear the SAM for at least 9 consecutive days. SAM was used to record the number of strides/minute following each visit. A stride is the leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again (that is, a stride generally equals 2 steps). The maximum continuous 10-minute, 20-minute, 30-minute, and 60-minute total step counts were computed for each participant. For each day, an active period was defined as the first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: Ambulatory 007e population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e, and had sufficient baseline and on-treatment data in Study 007e to assess measure of interest, excluding participants who had lost all independent ambulation. 'Number analyzed'=participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
steps
  Baseline: 10-minute total step count: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline: 10-minute total step count | 34.603 (12.4886) | 32.863 (8.8533) | 35.256 (10.0379) | 34.241 (10.5911)
  Change at Week 60: 10-minute total step count: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60: 10-minute total step count | -1.140 (6.9584) | -0.607 (7.2946) | -2.372 (7.1735) | -1.384 (7.1170)
  Baseline: 20-minute total step count: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline: 20-minute total step count | 28.138 (11.0629) | 26.096 (7.9168) | 28.323 (9.3133) | 27.526 (9.5426)
  Change at Week 60: 20-minute total step count: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60: 20-minute total step count | -1.459 (6.7165) | -0.662 (6.2171) | -2.510 (6.4346) | -1.558 (6.4549)
  Baseline: 30-minute total step count: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline: 30-minute total step count | 24.222 (9.9576) | 22.205 (7.1045) | 24.498 (8.4938) | 23.648 (8.6306)
  Change at Week 60: 30-minute total step count: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60: 30-minute total step count | -1.400 (5.7605) | -0.450 (5.6811) | -2.457 (5.9579) | -1.452 (5.8110)
  Baseline: 60-minute total step count: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline: 60-minute total step count | 18.019 (7.8145) | 16.453 (5.6625) | 18.599 (6.9509) | 17.691 (6.8991)
  Change at Week 60: 60-minute total step count: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60: 60-minute total step count | -0.977 (3.7328) | -0.210 (4.7035) | -2.257 (5.1038) | -1.162 (4.5803)

8. Secondary Outcome: Change From Baseline in Percentage of Time During Active Period Spent at No Activity (0 Steps/Minute[Min]), Low Activity (Less Than or Equal to [≤]15 Steps/Min), Medium Activity (16-30 Steps/Min), and High Activity (Greater Than[>]30 Steps/Min) at Week 60
Description: SAM is a pedometer (worn on the ankle) that continuously records the number of steps per time interval. Participants were instructed to continue to wear SAM for at least 9 consecutive days. SAM was used to record number of strides/minute following each visit. A stride is leg motion that begins when the foot with SAM leaves the floor and ends when the same foot touches the floor again. Percentage of time during active periods spent at no activity (0 steps/min), low activity (≤15 steps/min), medium activity (16-30 steps/min), and high activity (>30 steps/min) were computed for each participant. For each day, an active period was defined as first time after 3:00 AM that >2 strides/minute were recorded to the last time prior to midnight that >2 strides/minute were recorded. Days were deleted on which such an active period was <50% of the mean active period across all days for that participant's visit.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
percentage of time
  Baseline: Time spent at no activity: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline: Time spent at no activity | 52.818 (14.4129) | 53.372 (12.2352) | 50.006 (12.5263) | 52.094 (13.1188)
  Change at Week 60: Time spent at no activity: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60: Time spent at no activity | -0.051 (8.1776) | 0.830 (11.2481) | 2.194 (7.8652) | 0.985 (9.1467)
  Baseline: Time spent at low activity: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline: Time spent at low activity | 30.677 (7.8531) | 31.170 (7.2431) | 32.393 (7.2426) | 31.392 (7.4462)
  Change at Week 60: Time spent at low activity: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60: Time spent at low activity | 1.270 (5.8178) | 1.172 (8.3050) | 0.252 (5.5885) | 0.896 (6.6058)
  Baseline: Time spent at medium activity: number analyzed (Participants) | 52 | 49 | 48 | 149
  Baseline: Time spent at medium activity | 10.248 (4.7620) | 10.119 (4.4344) | 10.983 (4.6049) | 10.442 (4.5901)
  Change at Week 60: Time spent at medium activity: number analyzed (Participants) | 41 | 38 | 40 | 119
  Change at Week 60: Time spent at medium activity | -0.542 (2.0960) | -1.356 (3.7830) | -0.965 (3.3763) | -0.944 (3.1392)
  Baseline: Time spent at high activity: number analyzed (Participants) | 51 | 49 | 48 | 148
  Baseline: Time spent at high activity | 6.404 (4.5938) | 5.370 (3.4243) | 6.673 (4.5847) | 6.149 (4.2476)
  Change at Week 60: Time spent at high activity: number analyzed (Participants) | 39 | 38 | 40 | 117
  Change at Week 60: Time spent at high activity | -0.643 (2.2656) | -0.520 (2.7196) | -1.506 (2.9904) | -0.898 (2.6913)

9. Secondary Outcome: Change From Baseline in Time to Stand From Supine Position at Week 60
Description: If the time taken to perform this test exceeded 30 seconds or if a participant could not perform this test due to disease progression, a value of 30 seconds was used. Change from baseline data has been reported.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
seconds
  Baseline | 13.736 (11.3353) | 11.796 (10.3544) | 12.398 (11.6010) | 12.666 (11.0678)
  Change at Week 60: number analyzed (Participants) | 49 | 47 | 48 | 144
  Change at Week 60 | 0.665 (3.0080) | -0.187 (4.6289) | 0.002 (4.6322) | 0.166 (4.1373)

10. Secondary Outcome: Change From Baseline in Time to Walk/Run 10 Meters at Week 60
Description: as for outcome 9
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
seconds
  Baseline | 8.143 (5.1475) | 6.986 (2.9995) | 6.967 (3.5789) | 7.384 (4.0530)
  Change at Week 60: number analyzed (Participants) | 49 | 47 | 48 | 144
  Change at Week 60 | 1.441 (4.4822) | 0.547 (2.2058) | 0.758 (2.6862) | 0.922 (3.2905)

11. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs at Week 60
Description: as for outcome 9
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
seconds
  Baseline | 9.077 (9.2543) | 6.738 (6.4069) | 8.071 (9.2057) | 7.984 (8.4076)
  Change at Week 60: number analyzed (Participants) | 49 | 47 | 48 | 144
  Change at Week 60 | 0.831 (2.4664) | 0.696 (4.0707) | 0.194 (2.5268) | 0.574 (3.0898)

12. Secondary Outcome: Change From Baseline in Time to Descend 4 Stairs at Week 60
Description: as for outcome 9
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
seconds
  Baseline | 7.685 (8.9934) | 5.638 (5.5635) | 6.641 (7.8591) | 6.675 (7.6319)
  Change at Week 60: number analyzed (Participants) | 49 | 47 | 48 | 144
  Change at Week 60 | 1.167 (4.7624) | 0.626 (5.2567) | -0.648 (4.9202) | 0.385 (5.0045)

13. Secondary Outcome: Change From Baseline in Heart Rate Before, During, and After Each 6MWD Test at Week 60, as Assessed by Heart Rate Monitoring With the Polar® RS400
Description: The heart rate was measured with a Polar RS400 heart rate monitor, which consists of a transmitter strap worn around the chest and a wristwatch receiver. The monitor produces a digital text file with 1 value per minute that represents the mean heart rate for that minute. Mean heart rates values were collected prior to, during, and after the 6MWT. The participant rested for 5 minutes in a sitting position prior to the 6MWT, and the mean heart rate for the last minute of this rest period was collected and documented as the resting heart rate. During the 6MWT, the mean heart rate was collected and documented as the active heart rate. After completing the 6MWT and resting for 3 minutes, the mean heart rate for 1 minute was collected and documented as the recovery heart rate.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 53 | 50 | 49 | 152
beats/minute
  Baseline: Resting heart rate: number analyzed (Participants) | 52 | 50 | 48 | 150
  Baseline: Resting heart rate | 105.3 (13.29) | 108.8 (10.71) | 103.7 (12.98) | 105.9 (12.48)
  Change at Week 60: Resting heart rate: number analyzed (Participants) | 45 | 46 | 43 | 134
  Change at Week 60: Resting heart rate | 4.0 (13.91) | 3.7 (10.11) | 4.8 (10.82) | 4.2 (11.65)
  Baseline: Active heart rate: number analyzed (Participants) | 52 | 48 | 48 | 148
  Baseline: Active heart rate | 138.7 (21.45) | 144.8 (14.55) | 138.6 (20.87) | 140.6 (19.36)
  Change at Week 60: Active heart rate: number analyzed (Participants) | 45 | 44 | 42 | 131
  Change at Week 60: Active heart rate | 1.6 (17.65) | 6.1 (15.45) | 2.4 (14.87) | 3.4 (16.07)
  Baseline: Recovery heart rate: number analyzed (Participants) | 52 | 48 | 48 | 148
  Baseline: Recovery heart rate | 110.0 (13.32) | 112.0 (12.17) | 109.4 (13.21) | 110.4 (12.88)
  Change at Week 60: Recovery heart rate: number analyzed (Participants) | 43 | 44 | 44 | 131
  Change at Week 60: Recovery heart rate | 2.1 (12.82) | 4.6 (12.57) | 2.3 (11.29) | 3.0 (12.20)

14. Secondary Outcome: Change From Baseline in Number of Digits Recalled Forwards and Backwards on Digit Span Task at Week 60
Description: Basic attention and working memory was measured using the digit span task. A series of digits (0-9) were presented to the child in an auditory format only. The task had 2 parts; in the forward condition, the child was requested to repeat back the digits in the order they were presented and in the backward condition, he was requested to reverse the order of presentation. A raw score of the total number of correct responses was converted to an age-scaled-score (z-score) by subtracting the corresponding mean and dividing by the corresponding standard deviation of a reference population for that age.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: Evaluable population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e, who had sufficient baseline and on-treatment data in Study 007e to assess the measure of interest. 'Number analyzed'=participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 58 | 56 | 56 | 170
z-score
  Baseline: Forward condition: number analyzed (Participants) | 56 | 54 | 51 | 161
  Baseline: Forward condition | 4.1 (2.97) | 3.6 (2.54) | 3.2 (2.21) | 3.6 (2.61)
  Change at Week 60: Forward condition: number analyzed (Participants) | 52 | 51 | 51 | 154
  Change at Week 60: Forward condition | 0.0 (1.53) | 0.0 (1.19) | 0.0 (1.22) | 0.0 (1.32)
  Baseline: Backward condition: number analyzed (Participants) | 56 | 54 | 51 | 161
  Baseline: Backward condition | 1.4 (0.98) | 1.3 (0.82) | 1.2 (0.66) | 1.3 (0.84)
  Change at Week 60: Backward condition: number analyzed (Participants) | 49 | 51 | 49 | 149
  Change at Week 60: Backward condition | 0.1 (0.86) | -0.1 (0.66) | 0.0 (0.58) | 0.0 (0.71)

15. Secondary Outcome: Change From Baseline in Participant- Reported Health-Related Quality of Life (HRQL) as Measured by the Pediatric Quality of Life Inventory (PedsQL) Physical, Emotional, Social, and School Functioning Domain Scores at Week 60
Description: HRQL was measured via the PedsQL. The generic core module (including physical, emotional, social and school functioning scales) comprises 23 questions and the fatigue-specific module (including general fatigue, sleep/rest fatigue, and cognitive fatigue scales) comprises an additional 18 questions. The PedsQL was completed by both the participant and/or a parent/caregiver. Examples of items in each of the generic core module scales include: "It is hard for me to run"; "I feel sad or blue"; "I cannot do things that other kids my age can do;" and "It is hard to pay attention in class." Each of the generic core module items was scored on a 5-point Likert response scale from 0 (never a problem) to 4 (almost always a problem). Scores were transformed on a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating better health-related quality of life. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 60.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 58 | 56 | 56 | 170
units on a scale
  Baseline: Physical functioning score: number analyzed (Participants) | 54 | 54 | 49 | 157
  Baseline: Physical functioning score | 63.8145 (24.46918) | 63.3019 (22.72039) | 60.4865 (22.33484) | 62.5995 (23.11654)
  Change at Week 60: Physical functioning score: number analyzed (Participants) | 50 | 47 | 49 | 146
  Change at Week 60: Physical functioning score | -0.5982 (14.91137) | -1.2538 (14.60384) | 1.2755 (19.01169) | -0.1804 (16.23570)
  Baseline: Emotional functioning score: number analyzed (Participants) | 54 | 54 | 49 | 157
  Baseline: Emotional functioning score | 76.852 (21.1530) | 73.241 (20.1681) | 73.265 (22.2568) | 74.490 (21.1086)
  Change at Week 60: Emotional functioning score: number analyzed (Participants) | 50 | 47 | 49 | 146
  Change at Week 60: Emotional functioning score | -1.675 (13.6361) | 2.128 (14.9181) | -0.995 (13.1621) | -0.223 (13.9106)
  Baseline: Social functioning score: number analyzed (Participants) | 54 | 54 | 50 | 158
  Baseline: Social functioning score | 72.5000 (21.60429) | 68.6111 (21.37748) | 71.3000 (21.32858) | 70.7911 (21.36670)
  Change at Week 60: Social functioning score: number analyzed (Participants) | 50 | 47 | 50 | 147
  Change at Week 60: Social functioning score | -2.2000 (13.48317) | 0.8511 (17.36185) | 0.3500 (15.15237) | -0.3571 (15.32468)
  Baseline: School functioning score: number analyzed (Participants) | 52 | 54 | 48 | 154
  Baseline: School functioning score | 72.019 (20.7756) | 71.111 (18.2918) | 69.063 (20.3861) | 70.779 (19.7213)
  Change at Week 60: School functioning score: number analyzed (Participants) | 47 | 46 | 47 | 140
  Change at Week 60: School functioning score | -1.064 (16.5153) | -1.630 (17.7029) | 1.809 (16.9214) | -0.286 (16.9931)

16. Secondary Outcome: Change From Baseline in Parent/Caregiver- Reported HRQL as Measured by the PedsQL Physical, Emotional, Social, and School Functioning Domain Scores at Week 60
Description: HRQL was measured via the PedsQL. The generic core module (including physical, emotional, social and school functioning scales) comprises 23 questions and the fatigue-specific module (including general fatigue, sleep/rest fatigue, and cognitive fatigue scales) comprises an additional 18 questions. The PedsQL was completed by both the participant and/or a parent/caregiver. Examples of items in each of the generic core module scales include: "It is hard for me to run"; "I feel sad or blue"; "I cannot do things that other kids my age can do;" and "It is hard to pay attention in class." Each of the generic core module items was scored on a 5-point likert response scale from 0 (never a problem) to 4 (almost always a problem). Scores were transformed on a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating better health-related quality of life. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 48.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 58 | 56 | 56 | 170
units on a scale
  Baseline: Physical functioning score: number analyzed (Participants) | 57 | 55 | 56 | 168
  Baseline: Physical functioning score | 56.8217 (23.80718) | 52.5162 (20.02845) | 52.6307 (24.35727) | 54.0152 (22.78661)
  Change at Week 60: Physical functioning score: number analyzed (Participants) | 52 | 49 | 54 | 155
  Change at Week 60: Physical functioning score | -0.8499 (12.75478) | -1.1662 (13.27447) | -0.1736 (14.75049) | -0.7143 (13.55924)
  Baseline: Emotional functioning score: number analyzed (Participants) | 57 | 55 | 56 | 168
  Baseline: Emotional functioning score | 74.7368 (17.73870) | 72.5455 (16.04025) | 68.2813 (22.05309) | 71.8676 (18.87211)
  Change at Week 60: Emotional functioning score: number analyzed (Participants) | 52 | 49 | 54 | 155
  Change at Week 60: Emotional functioning score | -1.9231 (11.11289) | -0.3061 (13.32323) | -1.9213 (16.86642) | -1.4113 (13.95342)
  Baseline: Social functioning score: number analyzed (Participants) | 57 | 55 | 56 | 168
  Baseline: Social functioning score | 61.9518 (19.07606) | 61.6136 (15.44605) | 59.7545 (21.34593) | 61.1086 (18.71300)
  Change at Week 60: Social functioning score: number analyzed (Participants) | 52 | 49 | 54 | 155
  Change at Week 60: Social functioning score | 1.5144 (13.03356) | -0.7908 (11.34994) | 0.3472 (12.76238) | 0.3790 (12.38287)
  Baseline: School functioning score: number analyzed (Participants) | 56 | 55 | 55 | 166
  Baseline: School functioning score | 68.6607 (16.05363) | 64.0000 (15.07389) | 65.9091 (18.20894) | 66.2048 (16.50694)
  Change at Week 60: School functioning score: number analyzed (Participants) | 50 | 48 | 53 | 151
  Change at Week 60: School functioning score | 0.8000 (9.60230) | 1.6667 (10.93177) | -1.0377 (12.60946) | 0.4305 (11.13464)

17. Secondary Outcome: Change From Baseline in Participant-Reported HRQL as Measured by the Total Fatigue Scale Score at Week 60
Description: HRQL was measured via the PedsQL. The fatigue-specific module (including general fatigue, sleep/rest fatigue, and cognitive fatigue scales) comprises an additional 18 questions. PedsQL was completed by both the participant and/or a parent/caregiver. Fatigue-specific module obtains information relating to items such as: "I feel too tired to do things that I like to do"; "I spend a lot of time in bed"; and "I have trouble remembering more than one thing at a time;" Each of the fatigue-specific module items was scored on a 5-point Likert response scale from 0 (never a problem) to 4 (almost always a problem). Scores were transformed on a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating less fatigue. Total score was the sum of all items over the number of items answered on all scales. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 60.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: Evaluable population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e, who had sufficient baseline and on-treatment data in Study 007e to assess the measure of interest. 'Number analyzed'=participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 58 | 56 | 56 | 170
units on a scale
  Baseline: number analyzed (Participants) | 55 | 53 | 51 | 159
  Baseline | 76.7968 (18.31310) | 72.7833 (20.95237) | 72.5947 (17.32956) | 74.1111 (18.92041)
  Change at Week 60: number analyzed (Participants) | 50 | 46 | 49 | 145
  Change at Week 60 | -2.0484 (9.77928) | 0.3650 (15.94374) | -1.8049 (11.12724) | -1.2005 (12.42615)

18. Secondary Outcome: Change From Baseline in Parent/Caregiver-Reported HRQL as Measured by the Total Fatigue Scale Score at Week 60
Description: HRQL was measured via the PedsQL. The fatigue-specific module (including general fatigue, sleep/rest fatigue, and cognitive fatigue scales) comprises an additional 18 questions. The PedsQL was completed by both the participant and/or a parent/caregiver. Fatigue-specific module obtains information relating to items such as: "I feel too tired to do things that I like to do"; "I spend a lot of time in bed"; and "I have trouble remembering more than one thing at a time;" Each of the fatigue-specific module items was scored on a 5-point likert response scale from 0 (never a problem) to 4 (almost always a problem). Scores were transformed on a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating less fatigue. Total score was the sum of all items over the number of items answered on all scales. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 60.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 58 | 56 | 56 | 170
units on a scale
  Baseline: number analyzed (Participants) | 56 | 53 | 56 | 165
  Baseline | 75.7864 (13.88014) | 71.6596 (12.78488) | 71.1062 (13.62739) | 72.8724 (13.53355)
  Change at Week 60: number analyzed (Participants) | 53 | 46 | 54 | 153
  Change at Week 60 | -0.3272 (6.64218) | 1.2219 (10.11693) | 0.2269 (8.55130) | 0.3341 (8.44319)

19. Secondary Outcome: Change From Baseline in Participant and Parent/Caregiver Reported Activities of Daily Living of Participants Who Were Unable to Complete the 6MWT (Nonambulatory Participants), as Measured by the Egen Klassifikation (EK) Scale at Week 60
Description: Activities of daily living were measured using the EK scale in all participants who were unable to complete the 6MWT at Screening/Baseline on Day 1. The EK scale is an ordinal scale ranging from 0 to 30 points where 0 represents the highest level of independent function and 30 the lowest. The scale consists of 10 categories (each scored 0 to 3), involving different functional domains including 1) ability to use wheelchair, 2) ability to transfer from wheelchair, 3) ability to stand, 4) ability to balance in the wheelchair, 5) ability to move the arms, 6) ability to use the hands and arms when eating, 7) ability to turn in bed, 8) ability to cough, 9) ability to speak, and 10) physical well-being. The administration of the EK scale consisted of an interview of the participant to capture how he performed the tasks of daily life (as described by Categories 1 to 9) and how he perceived his well-being (as described by Category 10).
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: Non-Ambulatory 007e population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e, and who had lost all independent ambulation prior to entering Study 007e. 'Number analyzed'=participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 5 | 4 | 6 | 15
units on a scale
  Baseline: number analyzed (Participants) | 4 | 4 | 5 | 13
  Baseline | 3.0 (2.00) | 4.3 (0.50) | 3.2 (1.92) | 3.5 (1.61)
  Change at Week 60: number analyzed (Participants) | 4 | 4 | 5 | 13
  Change at Week 60 | 1.5 (0.58) | 0.8 (1.26) | -0.8 (1.48) | 0.4 (1.50)

20. Secondary Outcome: Change From Baseline in Parent/Caregiver-Reported Treatment Satisfaction Questionnaire for Medication (TSQM) Score at Week 60
Description: TSQM consisted of 14 questions about treatment satisfaction with drug in 4 domains: Effectiveness (Questions 1-3 scored as 1 [extremely dissatisfied] to 7 [extremely satisfied]), Side Effects (question 4 scored as 0 [no] or 1 [yes]; question 5 scored as 1 [extremely bothersome] to 5 [not at all bothersome]; questions 6 - 8 scored as 1 [a great deal] to 5 [not at all]), Convenience (questions 9 and 10 scored as 1 [extremely difficult] to 7 [extremely easy]; question 11 scored as 1 [extremely inconvenient] to 5 [extremely convenient]) and Global Satisfaction (question 12 scored as 1 [not at all confident] to 7 [extremely confident]; question 13 scored as 1 [not at all certain] to 5 [extremely certain]; question 14 scored as 1 [extremely dissatisfied] to 5 [extremely satisfied]). The scores of each of the domains were added together and an algorithm was used to create a score of 0 to 100, with higher scores indicating better treatment satisfaction.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 58 | 56 | 56 | 170
units on a scale
  Baseline: Effectiveness score: number analyzed (Participants) | 53 | 54 | 52 | 159
  Baseline: Effectiveness score | 56.8134 (26.72451) | 53.8580 (21.53292) | 50.4274 (22.96804) | 53.7212 (23.82541)
  Change at Week 60: Effectiveness score: number analyzed (Participants) | 50 | 46 | 50 | 146
  Change at Week 60: Effectiveness score | 2.7778 (15.52191) | 5.6159 (19.53233) | 1.7778 (14.99307) | 3.3295 (16.68460)
  Baseline: Side-effects score: number analyzed (Participants) | 55 | 55 | 54 | 164
  Baseline: Side-effects score | 96.8182 (10.81681) | 97.7273 (7.64176) | 96.8364 (8.94695) | 97.1291 (9.18246)
  Change at Week 60: Side-effects score: number analyzed (Participants) | 51 | 47 | 48 | 146
  Change at Week 60: Side-effects score | 0.7353 (12.16084) | -1.0638 (7.74500) | -1.2587 (10.84441) | -0.4994 (10.43907)
  Baseline: Convenience score: number analyzed (Participants) | 57 | 55 | 54 | 166
  Baseline: Convenience score | 57.4074 (16.10609) | 57.9798 (19.05889) | 60.5967 (16.65858) | 58.6345 (17.26216)
  Change at Week 60: Convenience score: number analyzed (Participants) | 53 | 47 | 50 | 150
  Change at Week 60: Convenience score | 0.8386 (12.39372) | -1.6548 (11.75175) | 1.3333 (9.80472) | 0.2222 (11.38059)
  Baseline: Global satisfaction score: number analyzed (Participants) | 55 | 55 | 54 | 164
  Baseline: Global satisfaction score | 61.4286 (25.95857) | 60.4870 (23.30835) | 56.7791 (21.25768) | 59.5819 (23.54109)
  Change at Week 60: Global satisfaction score: number analyzed (Participants) | 53 | 47 | 50 | 150
  Change at Week 60: Global satisfaction score | -0.2695 (13.57882) | 1.2538 (15.30213) | -0.4643 (14.78188) | 0.1429 (14.45922)

21. Secondary Outcome: Change From Baseline in Serum Concentration of Creatine Kinase (CK) at Week 60
Description: Blood samples collected for chemistry assays were used to quantify serum CK concentrations. Serum CK was assessed as a potential biomarker for muscle fragility, with a reduction in serum CK considered to be a positive outcome.
Time Frame: Baseline (Week 48 of Study 007), Week 60
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units/liter (U/L)
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 58 | 56 | 56 | 170
units/liter (U/L)
  Baseline: number analyzed (Participants) | 57 | 56 | 54 | 167
  Baseline | 9163.1 (5542.80) | 10009.1 (5828.26) | 9150.7 (5657.67) | 9442.8 (5656.99)
  Change at Week 60: number analyzed (Participants) | 49 | 51 | 53 | 153
  Change at Week 60 | -455.1 (4962.00) | -520.5 (6164.96) | -334.3 (4810.45) | -435.1 (5310.37)

22. Secondary Outcome: Study Drug Compliance
Description: Study drug compliance was assessed by participant daily diary and quantification of used and unused study drug. Compliance was assessed in terms of the percentage of drug actually taken relative to the amount that should have been taken during the study.
Time Frame: Baseline (Week 48 of Study 007) to Week 96
Population: As-treated population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e.
Measure: Median (Full Range); unit: percentage of drug
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 59 | 57 | 57 | 173
percentage of drug | 0.00 [0.0 to 45.1] | 0.00 [0.0 to 10.5] | 0.00 [0.0 to 36.1] | 0.00 [0.0 to 45.1]

23. Secondary Outcome: Trough Ataluren Plasma Concentration
Description: Plasma samples for the determination of ataluren concentrations were analyzed at the bioanalytical laboratory for ataluren parent drug using a validated high performance liquid chromatography with tandem mass spectrometry (HPLC/MS-MS) method with a lower limit of quantitation (LLOQ) of 0.5 micrograms/millilitre (mcg/mL). Values below the LLOQ were set to 0.
Time Frame: Pre-morning dose (0 hour) at Baseline (Week 48 of 007 study), Weeks 54, 60, 72, 84, and 96
Population: As-treated population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e. 'Number analyzed'=participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Number analyzed (Participants) | 59 | 57 | 57 | 173
mcg/mL
  Week 48: number analyzed (Participants) | 58 | 57 | 57 | 172
  Week 48 | 12.656 (10.8951) | 4.541 (3.4381) | 0.000 (0.0000) | 5.773 (8.4333)
  Week 54: number analyzed (Participants) | 58 | 57 | 56 | 171
  Week 54 | 10.801 (8.4858) | 13.941 (14.5222) | 11.564 (9.3312) | 12.097 (11.1172)
  Week 60: number analyzed (Participants) | 55 | 54 | 56 | 165
  Week 60 | 11.547 (9.6034) | 13.830 (11.9096) | 13.302 (9.4765) | 12.890 (10.3574)
  Week 72: number analyzed (Participants) | 25 | 21 | 19 | 65
  Week 72 | 12.279 (10.5894) | 13.930 (10.6393) | 10.948 (6.3465) | 12.424 (9.4948)
  Week 84: number analyzed (Participants) | 6 | 7 | 5 | 18
  Week 84 | 15.232 (8.8909) | 14.773 (10.4404) | 11.082 (14.6331) | 13.901 (10.7415)
  Week 96: number analyzed (Participants) | 1 | 2 | 0 | 3
  Week 96 | 8.430 | 5.685 (2.7648) |  | 6.600 (2.5167)

ADVERSE EVENTS:
Time Frame: Baseline (Week 48 of Study 007) up to Week 102
Description: As-treated population included all participants who completed Study 007 and received ≥1 dose of ataluren in Study 007e.
Arm/Group | High-Dose Ataluren/High-Dose Ataluren | Low-Dose Ataluren/High-Dose Ataluren | Placebo/High-Dose Ataluren | Overall Participants: High-Dose Ataluren
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/57 | 2/57 | 3/173
Other Adverse Events (participants affected / at risk) | 53/59 | 51/57 | 51/57 | 155/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Dose Ataluren/High-Dose Ataluren (N=59) | Low-Dose Ataluren/High-Dose Ataluren (N=57) | Placebo/High-Dose Ataluren (N=57) | Overall Participants: High-Dose Ataluren (N=173)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Ataluren/High-Dose Ataluren (N=59) | Low-Dose Ataluren/High-Dose Ataluren (N=57) | Placebo/High-Dose Ataluren (N=57) | Overall Participants: High-Dose Ataluren (N=173)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dilatation ventricular (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Kidney malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (5)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Myopia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (16) | 12 (23) | 20 (33) | 43 (72)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 11 (13) | 6 (8) | 20 (25)
Abdominal pain (Gastrointestinal disorders) | 6 (10) | 4 (4) | 6 (7) | 16 (21)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 9 (11) | 4 (5) | 15 (18)
Flatulence (Gastrointestinal disorders) | 7 (7) | 4 (4) | 3 (3) | 14 (14)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (4) | 3 (3) | 11 (12)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 4 (5)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disease progression (General disorders) | 9 (9) | 7 (7) | 3 (3) | 19 (19)
Asthenia (General disorders) | 2 (3) | 5 (5) | 2 (2) | 9 (10)
Gait disturbance (General disorders) | 4 (4) | 3 (3) | 2 (2) | 9 (9)
Pyrexia (General disorders) | 4 (4) | 2 (3) | 3 (4) | 9 (11)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 7 (7) | 5 (5) | 6 (6) | 18 (18)
Nasopharyngitis (Infections and infestations) | 3 (4) | 8 (10) | 5 (5) | 16 (19)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 3 (4) | 5 (5) | 14 (17)
Ear infection (Infections and infestations) | 2 (3) | 2 (2) | 4 (5) | 8 (10)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (2) | 3 (3) | 7 (8)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 3 (4) | 5 (6)
Otitis media (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 5 (6)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (4) | 3 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 1 (3) | 2 (4)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 5 (5) | 4 (4) | 14 (15)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0) | 3 (4)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (11) | 3 (3) | 4 (7) | 11 (21)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 2 (2) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8) | 4 (4) | 1 (1) | 10 (14)
Joint contracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (8) | 1 (1) | 9 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0) | 7 (7)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 6 (6)
Lordosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 1 (1) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (5) | 1 (1) | 6 (7)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (48) | 15 (48) | 14 (17) | 34 (113)
Migraine (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Areflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Frustration (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oppositional defiant disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enuresis (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 6 (6)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Kidney enlargement (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin chapped (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 6 (6) | 13 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2) | 1 (1) | 7 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 0 (0) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was prematurely terminated by Sponsor per Data Monitoring Committee (DMC) recommendation to discontinue ongoing studies of high-dose ataluren in nmDBMD due to lack of efficacy for the high-dose ataluren.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.